CLINICAL TRIAL: NCT00347490
Title: Efficacy and Safety in Hemodialysis With Enoxaparine
Brief Title: HENOX: Enoxaparine in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENOXA_L_00821
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Enoxaparin

INTERVENTIONS:
Drug: Enoxaparine

SUMMARY:
Primary objective:

To assess clinical efficacy of single bolus anticoagulation with Enoxaparin in chronic hemodialysis

Secondary objective:

To assess safety and tolerability by the number of spontaneously reported adverse events by patients

ELIGIBILITY:
Inclusion Criteria:

* End stage renal failure requiring maintenance hemodialysis at least twice a week
* Has arterio-venous fistula or arterio-venous graft in upper extremities which can apply to blood flow > or = 250ml/min as a vascular access for hemodialysis.
* Stable hemodialysis prescription at least 1 month before enrollment
* UFH (Unfractionated Heparin) was prescribed as an anticoagulant in the previous hemodialysis prescription
* No sign of active infection .
* Absence of recent cardiovascular complication such as myocardial infarction, DVT (Deep Venous Thrombosis), arterial occlusion, pulmonary embolism, cerebrovascular disease in previous 3 months.

Exclusion Criteria:

* Women who are breastfeeding, pregnant or of childbearing age and not using medically acceptable effective contraception
* Patients with any evidence of an active bleeding disorder
* Contraindication to anticoagulation:

  * Prior history of cerebral hemorrhage at any time
  * Coagulopathy (acquired or inherited)
  * Recent surgery
  * Major surgery such as neurosurgery within the past 3 months
  * Minor surgery such as intraocular surgery within 1 month.
  * Uncontrolled predialytic arterial hypertension (systolic BP > 200 mmHg or diastolic BP > 110 mmHg) at 2 successive readings
  * Impaired hemostasis i.e., known or suspected coagulopathy (acquired or inherited): baseline platelet count <100,000/mm3 in patients without baseline diagnosis of active cancer and undergoing chemotherapy treatment (for patients with diagnosis of cancer and undergoing chemotherapy, baseline platelet count >70,000/mm3); aPTT (activated Partial Thromboplastin Time) 1.5X the laboratory upper limit of normal; or international normalized ratio (INR) >1.5
* Indication for thrombolytic therapy such as ischemic heart disease, ischemic stroke.
* Need for a curative treatment of anticoagulant therapy(DVT ,pulmonary embolism, ischemic heart disease)
* Patients treated with oral anticoagulant therapy within 72 hours prior to inclusion
* Patients who have had spinal or epidural analgesia or lumbar puncture within the preceding 24 hours
* Abnormal liver enzyme and total bilirubin within 2 weeks (SGPT, SGOT, total bilirubin above 2 times of Upper normal limit)
* Known hypersensitivity to heparin or LMWH (Low Molecular Weight Heparin), or pork derived products
* History of documented episode of heparin or LMWH induced thrombocytopenia and/or thrombosis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Rate of fibrin / clot formation in dialyser and line grade in 10-point scale

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sompob Paibulsirijit, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bangkok, Thailand